CLINICAL TRIAL: NCT04628936
Title: An Open-label Extension to the Phase 2 Randomized, Double-blind, Placebo-controlled, Crossover Multicenter Study to Evaluate the Safety and Efficacy of KZR-616 in the Treatment of Patients With Active Polymyositis or Dermatomyositis
Brief Title: Open-label Extension to the Phase 2 Crossover Study (PRESIDIO) Evaluating KZR-616 in Patients With PM and DM.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kezar Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KZR-616-003E
Record Dates: First submitted 2020-11-02; First posted 2020-11-16 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Polymyositis; Dermatomyositis
Keywords: Myositis; Idiopathic inflammatory myopathies; Polymyositis; Dermatomyositis; Musculoskeletal Diseases; Muscular Diseases
MeSH Terms: conditions — Polymyositis; Dermatomyositis; Myositis; Musculoskeletal Diseases; Muscular Diseases | interventions — KZR-616

STUDY DESIGN:
Intervention Model Description: All patients received a SC injection of 30 mg KZR-616 at Visit 1 (Day 1), followed by weekly SC injections of 45 mg KZR-616 up to a maximum of 96 weeks. Study drug administration ended for all patients when the last patient enrolled completed 48 weeks of dosing.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KZR-616 45 mg + standard therapy (open-label) (Experimental): All patients received a SC injection of 30 mg KZR-616 at Visit 1 (Day 1), followed by weekly SC injections of 45 mg KZR-616 up to a maximum of 96 weeks. Study drug administration ended for all patients in Study KZR-616-003E when the last patient enrolled completed 48 weeks of dosing.
  Interventions: Drug: KZR-616

INTERVENTIONS:
Drug: KZR-616 — Subcutaneous 30 mg for 1 week, then 45 mg weekly
  Other Names: KZR-616 Lyophile; zetomipzomib

SUMMARY:
This was an open-label study to evaluate the long-term efficacy and safety of KZR-616 in patients with active polymyositis (PM) or dermatomyositis (DM) who completed the double-blind treatment period of Study KZR-616-003, up to and including the Week 32 Visit, prior to the first dose of open-label KZR-616.

DETAILED DESCRIPTION:
This was an open-label study to evaluate the long-term efficacy and safety of KZR-616 in patients with active polymyositis or dermatomyositis who completed the double-blind treatment period of Study KZR-616-003 (NCT04033926), up to and including the Week 32 Visit, prior to the first dose of open-label KZR-616.

Patients were evaluated for eligibility according to the entry criteria at, or within 8 weeks after, the Week 32 Visit (ie, the End of Treatment [EOT] Visit [Visit 34]) of Study KZR-616-003.

All patients received a subcutaneous (SC) injection of 30 mg KZR-616 at Visit 1 (Day 1), followed by weekly SC injections of 45 mg KZR-616 up to a maximum of 96 weeks. Study drug administration ended for all patients in Study KZR-616-003E when the last patient enrolled completed 48 weeks of dosing. Patients had a final follow-up visit 12 weeks after their last dose of KZR-616 (End of Study [EOS] Visit), for a maximum potential length of participation of 108 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Must have successfully completed Study KZR-616-003 through Week 32, including the Week 32 Visit assessments
* Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test prior to the first dose of KZR-616 in KZR-616-003E, and must agree to continue to use a highly effective method of birth control until completion of the study.
* Male patients must continue to use an effective contraception method for 1 week following their last dose of KZR-616 or be congenitally or surgically sterile.

Exclusion Criteria:

* Has participated in any clinical study other than KZR-616-003 between the Week 32 Visit of Study KZR-616-003 and the first study visit of KZR-616-003E, if they are not on the same calendar day.
* Are females who are breastfeeding or who plan to become pregnant during the study, or who are actively trying to conceive at the time of signing of the informed consent form.
* Have hypersensitivity to KZR-616 or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kezar Study Director, Study Director — Kezar Life Sciences, Inc.
Locations (10):
- United States (9):
  - KZR Research Site, Beverly Hills, California
  - KZR Research Site, Orange, California
  - KZR Research Site, Miami, Florida
  - KZR Research Site, Kansas City, Kansas
  - KZR Research Site, Baltimore, Maryland
  - KZR Research Site, Ann Arbor, Michigan
  - KZR Research Site, Duncansville, Pennsylvania
  - KZR Research Site, Pittsburgh, Pennsylvania
  - KZR Research Site, Austin, Texas
- KZR Research Site, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Kezar Life Sciences, Inc. corporate website — https://www.kezarlifesciences.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- KZR-616 45 mg + Standard Therapy (Open-label): All patients received SC injections of KZR-616 once weekly (QW) at doses of 30 mg on day 1 and 45 mg thereafter for up to 96 weeks. Study drug administration ended when the last enrolled patient completed 48 weeks of dosing in the OLE. Patients had an end of study visit 12 weeks after the last dose of KZR-616.
  KZR-616: zetomipzomib subcutaneous injection
Period: Overall Study
Arm/Group | KZR-616 45 mg + Standard Therapy (Open-label)
Started | 18
Completed | 8
Not Completed | 10

BASELINE CHARACTERISTICS:
Groups:
- KZR-616 45 mg + Standard Therapy (Open-label): All patients received SC injections of KZR-616 QW at doses of 30 mg on day 1 and 45 mg thereafter for up to 96 weeks. Study drug administration ended when the last enrolled patient completed 48 weeks of dosing in the OLE. Patients had an end of study visit 12 weeks after the last dose of KZR-616.
  KZR-616: zetomipzomib subcutaneous injection
Arm/Group | KZR-616 45 mg + Standard Therapy (Open-label)
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Improvement Score (TIS) at OLE Week 48
Description: The mean Total Improvement Score (TIS) at OLE Week 48, which ranges from 0 to 100 [low of 0 to high of 100, where higher scores are better]. The timeframe of 48 weeks was selected because it represented the maximum timeframe of dosing for the last patient enrolled as the study drug administration ended when the last patient enrolled completed 48 weeks of dosing.
Time Frame: 48 weeks
Population: Nine (9) patients were enrolled in the OLE study at Week 48.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | KZR-616 45 mg + Standard Therapy (Open-label)
Number analyzed (Participants) | 9
score on a scale | 36.4 (23.2)

ADVERSE EVENTS:
Time Frame: Up to 108 weeks
Description: Anticipated fluctuations of pre-existing conditions, including the disease under study, that do not represent a clinically significant exacerbation or worsening were not considered adverse events for this study.
Arm/Group | KZR-616 45 mg + Standard Therapy (Open-label)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KZR-616 45 mg + Standard Therapy (Open-label) (N=18)
Wellens' syndrome (Cardiac disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KZR-616 45 mg + Standard Therapy (Open-label) (N=18)
Angina pectoris (Cardiac disorders) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (6)
Diverticulum intestinal (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (31)
Vomiting (Gastrointestinal disorders) | 4 (8)
Asthenia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 4 (14)
Fatigue (General disorders) | 3 (41)
Influenza like illness (General disorders) | 1 (1)
Infusion site reaction (General disorders) | 1 (1)
Injection site bruising (General disorders) | 3 (47)
Injection site erythema (General disorders) | 4 (98)
Injection site exfoliation (General disorders) | 1 (2)
Injection site induration (General disorders) | 3 (6)
Injection site inflammation (General disorders) | 1 (1)
Injection site irritation (General disorders) | 1 (2)
Injection site pain (General disorders) | 1 (10)
Injection site pruritus (General disorders) | 2 (24)
Injection site rash (General disorders) | 1 (1)
Injection site reaction (General disorders) | 8 (177)
Injection site swelling (General disorders) | 2 (33)
Injection site urticaria (General disorders) | 1 (1)
Injection site vesicles (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pain (General disorders) | 5 (38)
Pyrexia (General disorders) | 5 (18)
Vaccination site pain (General disorders) | 1 (1)
Biliary dilatation (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (3)
Adenovirus infection (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)
Administration related reaction (Injury, poisoning and procedural complications) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (2)
Post vaccination syndrome (Injury, poisoning and procedural complications) | 2 (4)
Underdose (Injury, poisoning and procedural complications) | 1 (1)
Reticulocyte count increased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (9)
Migraine (Nervous system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (2)
Ureterolithiasis (Renal and urinary disorders) | 1 (2)
Menopausal symptoms (Reproductive system and breast disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (10)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall have the right to publish or present their own data resulting from the Study ("Publication") upon the earlier of: (a) the date following a multicenter publication coordinated by Sponsor regarding the Protocol; (b) 12 months after completion of the Protocol by all sites; or (c) the date after submission of the Study Data by Sponsor to the FDA.

The PI must furnish Sponsor with a copy of any Publication at least 30 days in advance of the proposed submission or presentation date.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT04628936/Prot_SAP_000.pdf